CLINICAL TRIAL: NCT04307862
Title: A Phase II Multicenter, Randomized, Double Blind Study to Assess the Safety, Tolerability and Efficacy of Two Concentrations of ZEP-3Na Topical Cream (0.1% and 1%) Compared to Vehicle-control in Subjects With Mild to Moderate Atopic Dermatitis With an Open Label Extension of up to 2 Weeks Treatment With ZEP-3Na Topical Cream 1%
Brief Title: Safety, Tolerability and Efficacy of ZEP-3Na (0.1% or 1%) Compared to Placebo in Subjects With Mild to Moderate Atopic Dermatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shulov Innovate for Science Ltd. 2012 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZEP-003-IL
Record Dates: First submitted 2019-11-24; First posted 2020-03-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZEP-3Na 0.1% (Experimental): The ZEP-3Na 0.1% cream will be applied topically twice daily
  Interventions: Drug: ZEP-3Na 0.1%
- ZEP-3Na 1% (Experimental): The ZEP-3Na 1% cream will be applied topically twice daily
  Interventions: Drug: ZEP-3Na 1%
- Vehicle Control (Placebo Comparator): The Vehicle Control cream will be applied topically twice daily
  Interventions: Drug: Placebo Vehicle only

INTERVENTIONS:
Drug: ZEP-3Na 0.1% — The Investigational Product will be applied topically twice daily for up to 4 weeks in the double blind phase
  Arms: ZEP-3Na 0.1%
Drug: ZEP-3Na 1% — The Investigational Product will be applied topically twice daily for up to 4 weeks in the double blind phase, with optional 2 weeks of open label with ZEP-3Na 1%.
  Arms: ZEP-3Na 1%
Drug: Placebo Vehicle only — he Investigational Product will be applied topically twice daily for up to 4 weeks in the double blind phase
  Arms: Vehicle Control

SUMMARY:
This is a phase II, double blind study with ZEP-3NA 0.1% or 1% vs. vehicle-control in subjects with mild to moderate Atopic Dermatitis. The IP (Investigational Product) will be administered topically twice daily for 4 weeks in the double blind phase. patients that will reach the primary endpoint will have the opportunity for additional to two weeks of open label treatment with ZEP-3Na 1%.

The purpose of this study is to assess the safety, tolerability and efficacy of two concentrations of ZEP-3NA compared to vehicle-control.

DETAILED DESCRIPTION:
165 subjects, 5-75 years old with mild to moderate Atopic Dermatitis will be enrolled to the study.

The investigational product which is the synthetic analogue of the natural compound found in the rattle snake venom will be administered topically twice daily.

The duration of the study will be up to 11 weeks consisting of up to 3 weeks of screening, 4 weeks of double blind treatment, optional 2 weeks of open label treatment, followed by 2 weeks of follow-up.

Efficacy will be measured by IGA (Investigator Global Assessment, EASI (Eczema Area and Severity Index) and SCORAD (SCORing Atopic Dermatitis).

Lesions will be photographed throughout the study. Physical examination and vital signs will be measured during every visit. Patients will complete quality of life questionnaires, itching scale and diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 5 to 75 years old, inclusive.
2. Clinical diagnosis of Atopic Dermatitis (as defined by Hanifin and Rajka criteria).
3. Atopic Dermatitis should be present for at least three months with stable disease for ≥ 1 month prior to screening.
4. IGA score of 2 or 3 (mild or moderate) during screening and baseline.
5. Women of child bearing potential must have a negative urine pregnancy test at screening and use an adequate contraceptive method throughout the study. Women of child bearing potential is defined as any female who has experienced menarche and who has not undergone surgical sterilization (such as: hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 24 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. Adequate method of birth control is defined as one of the following: oral or injectable contraceptives, intrauterine device, contraceptive implants, tubal ligation, hysterectomy, or a double-barrier method (diaphragm with spermicidal foam or jelly, or a condom), abstinence or vasectomy. Males with partners of childbearing potential should inform them of their participation in this clinical study and use an adequate contraceptive method throughout the study.
6. Willing and able to comply with study instructions and commit to attending all visits.
7. The patient/parent/guardian has the ability to understand, agree to and sign the study Informed Consent Form prior to performing any study-related procedure. Adolescents age >16 to 18 years old should be willing and able to sign Assent Form.

Exclusion Criteria:

1. Unstable or actively infected atopic dermatitis.
2. Concomitant dermatologic (e.g. irritant contact dermatitis, allergic contact dermatitis, psoriasis, etc.) or other medical condition(s) which may interfere with the investigator's ability to evaluate the subject's response to study drug.
3. Patients with Atopic Dermatitis affecting only the scalp will be excluded from the study. In addition, patients with the scalp representing ≥ 25% of the affected area will be excluded as well.
4. Has received treatment two weeks prior to visit 2 (Day 1 of IP) with topical corticosteroids and/or topical immunosuppressive drugs or four weeks prior to visit 2 (Day 1 of IP) with systemic immunosuppressive drugs and/or corticosteroids or plans to receive treatment during the study timeframe with immunosuppressive drugs and/or corticosteroids (topical or systemic).
5. Use of Crisaborole two weeks prior to visit 2 (Day 1 of IP).
6. Prior use of Dupilumab.
7. Subjects who are using any concomitant medications that, in the investigator's opinion, could affect the subject's atopic dermatitis (e.g Antihistamines). Subjects using such medications and have been stable on treatment for at least one month prior to visit 2 (Day 1 of IP) and no changes to these medications are planned during study, may be included in the study, at the investigator's discretion.
8. Subject had UVA or UVB therapy two weeks prior to visit 2 (Day 1 of IP) or is due to have it during the study period.
9. Any vaccination in the last 30 days prior to the screening visit. However, due to COVID-19 pandemic, only 1st vaccination for COVID is not allowed during only 21 days prior to visit 2 (Day 1 of IP) and during the study. The 2nd vaccination onwards is allowed at all times.
10. Abnormal renal function (defined as serum creatinine >1.5xULN).
11. Abnormal liver function (defined as any transaminases >2xULN).
12. Clinically significant abnormalities as determined by the Investigator on the 12-lead ECG conducted at the screening visit (for adults only).
13. Subject has active or history of malignancy, except non melanomatous skin cancer cured by excision. Subjects with past malignancy who had completed therapy and are free of the disease for at least 5 years may be included in the study, at the investigator's discretion.
14. History of immunodeficiency syndrome (e.g. atypical rash morphology, severe bacterial, fungal or viral skin infections, etc).
15. Subjects who are receiving any investigational drug or who participated in a clinical trial with an investigational product within the last 30 days or 5-half-lives of the investigational product, whichever is longer.
16. History of any anaphylactic reaction or history or evidence of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis and atopic dermatitis).
17. Known hypersensitivity to any of the components of the study drug.
18. Known or suspected history of alcohol or drug abuse.
19. Subjects with a history of human immunodeficiency virus (HIV) as determined by medical history.
20. Pregnant or lactating women.
21. Any history which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2019-12-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
• Proportion of subjects with IGA 0 to 1 (on a 5-point scale) and a reduction from baseline of ≥2 points during up to 4 weeks of double blind treatment | Up to 4 weeks
  Lower score of IGA mean better outcome, higher score mean worse outcome

SECONDARY OUTCOMES:
• Proportion of subjects with IGA 0 to 1 (on a 5-point scale) and a reduction from baseline of ≥2 points during up to 4 weeks of double blind treatment and following additional up to 2 weeks of an open label extension with ZEP 3Na 1%, if applicable | Up to 6 weeks
  Lower score of IGA mean better outcome, higher score mean worse outcome
• Proportion of subjects with EASI-50 (≥50% improvement from baseline) at end of treatment visit (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
  Higher score mean better outcome, lower score mean worse outcome
• Percent change in EASI-50 score from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
  Higher score mean better outcome, lower score mean worse outcome
• Percent change from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable) in pruritus NRS. | Up to 6 weeks
  Lower score of NRS mean better outcome, higher score mean worse outcome
• Proportion of subjects with improvement (reduction) of pruritus NRS ≥3 points from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
  Lower score of NRS mean better outcome, higher score mean worse outcome
• Change from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable) in SCORAD. | Up to 6 weeks
  Lower score of SCORAD mean better outcome, higher score mean worse outcome
• Distribution of disease severity scores (eg, IGA, EASI, SCORAD) and their change from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
• Proportion of subjects who achieve reduction of IGA score by ≥1 from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
• Proportion of subjects who achieve reduction of IGA score by ≥2 from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
Time to ≥1 point improvement in IGA. | Up to 6 weeks
  Lower score mean better outcome, higher score mean worse outcome
• Time to > 2 points improvement in IGA. | Up to 6 weeks
  Lower score mean better outcome, higher score mean worse outcome
• Change from baseline to EoT (EoT of the double blind part and EoT of the open label part, if applicable) in DLQI. | Up to 6 weeks
• Incidence of skin infection treatment-emergent adverse events (TEAE) requiring systemic treatment from baseline through EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
• Incidence of treatment-emergent serious adverse events (TESAEs) from baseline through EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
• Incidence of TEAEs leading to treatment discontinuation from baseline through EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks
• Overall incidence of TEAEs through EoT (EoT of the double blind part and EoT of the open label part, if applicable). | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- Israel (10):
  - Ha'Emek MC, Afula
  - Barzilai MC, Ashkelon
  - Rambam MC, Haifa
  - Shaare Zedek MC, Jerusalem
  - Clalit Health Services, Kfar Saba
  - Prof. Shemer Clinic affiliated to Laniado MC, Netanya
  - Clalit Health Services, Petah Tikva
  - Clalit Health Services, Ramla
  - Kaplan MC, Rehovot
  - Tel-Aviv Sourasky MC, Tel Aviv